CLINICAL TRIAL: NCT03874806
Title: Pharmacokinetic Profile and Dermatomal Coverage of the Erector Spinae Plane Block: a Comparison of Bolus Dosing and Continuous Infusion
Brief Title: Pharmacokinetic Profile and Dermatomal Coverage of the Erector Spinae Plane Block
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Did not receive funding
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20014803
Record Dates: First submitted 2019-03-08; First posted 2019-03-14 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Pain, Postoperative; Pain, Chest
MeSH Terms: conditions — Pain, Postoperative; Chest Pain | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- single (Experimental): local anesthetic is delivered as a single bolus
  Interventions: Drug: Ropivacaine 0.25%-NaCl 0.9% Injectable Solution
- continuous (Active Comparator): local anesthetic is delivered as a continuous infusion
  Interventions: Drug: Ropivacaine 0.2%-NaCl 0.9% Injectable Solution

INTERVENTIONS:
Drug: Ropivacaine 0.25%-NaCl 0.9% Injectable Solution — 0.25% ropivacaine administered through a nerve catheter
  Arms: single
Drug: Ropivacaine 0.2%-NaCl 0.9% Injectable Solution — 0.2% ropivacaine administered through a nerve catheter
  Arms: continuous

SUMMARY:
The goals of this study are as follows:

1. to confirm the safe dosing of ropivacaine for the erector spinae plane block
2. develop a pharmacokinetic profile of the erector spinae plane block, which will help demonstrate how quickly and how closely toxic levels are reached when a routine dose of ropivacaine is given for this nerve block
3. assess numbness created by the erector spinae block when routine doses are administered

ELIGIBILITY:
Inclusion Criteria:

1. Participant's age is greater than 18 years
2. Participant is undergoing a primary coronary artery bypass grafting surgery or heart valve replacement that requires a midline sternotomy incision
3. Participant's surgery is being performed by Dr. Vig Kasirajan

Exclusion Criteria:

1. Diagnosis of cirrhosis, hepatitis, primary sclerosing cholangitis
2. Abnormal liver function tests demonstrated by lab results
3. Allergy to lidocaine, ropivacaine, or midazolam
4. Morbid obesity, defined as body mass index greater than 40
5. Existing skin neuropathy on the chest or back
6. Body weight less than 50 kg
7. Participant is not able to provide verbal feedback, such as when the participant develops altered mental status or requires prolonged mechanical ventilation and sedation
8. Participant remains intubated on post-operative day 1
9. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Cmax | 28 hours
  The maximum concentration of serum ropivacaine after pre-determined dose is delivered through the ESP nerve catheter
Tmax | 28 hours
  The time elapsed from initial ropivacaine administration to Cmax
Area of analgesia | 4 hours
  The area of numbness experienced in the chest wall; measured using a pinprick test and documented on a cartoon map showing a chest wall and dermatomal borders
Duration of analgesia | 4 hours
  The duration of numbness to the chest wall; start time will be when the local anesthetic bolus is given, and end time will be when the participant reports the resolution of chest wall numbness

CONTACTS AND LOCATIONS:
Overall Officials: Bryant Tran, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/06/NCT03874806/Prot_SAP_000.pdf